CLINICAL TRIAL: NCT02443662
Title: Interstitial Colloid Osmotic Pressure in Children With Fontan Circulation After Fontan Surgery
Brief Title: Colloid Osmotic Pressure in Patients With Fontan Circulation
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Marianne Indrebo, MD, Oslo University Hospital
Other Study IDs: 063.09f
Record Dates: First submitted 2015-05-04; First posted 2015-05-14 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Catheterization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Interstitial fluid. Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Catheterization — Routine catheterization during follow up.

SUMMARY:
Children born with univentricular heart will go through step surgery and end up with a Fontan circulation. A circulation with cause problems with body fluid balance.This project will evaluate changes in interstitial colloid osmotic pressure in patients 10 year after completion of a three step Fontan surgery. This project will evaluate whether increased micro vascular leakage and change in interstitial colloid osmotic pressure are present in patients after ten years with a Fontan circulation.

ELIGIBILITY:
Inclusion Criteria:

* Fontan circulation after completed Fontan surgery.
* Anesthesia during catheterization.

Exclusion Criteria:

* No consent

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who will have a cathererization during their routine check up 10 years after completion of Fontan surgery.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Interstitial colloid osmotic pressure | Ten years after completed Fontan surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Indrebø, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided